CLINICAL TRIAL: NCT05469087
Title: Prospective Cohort Primary Hyperparathyroidism
Brief Title: Cohort Primary Hyperparathyroidism
Acronym: CoHPT
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC15_0424
Record Dates: First submitted 2022-07-07; First posted 2022-07-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Primary Hyperparathyroidism
Keywords: Primary hyperparathyroidism; Parathyroidectomy
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
CoHPT is a prospective, monocentric, observational cohort including all patients diagnosed with primary hyperparathyroidism in Nantes University Hospital, aiming to study the outcomes associated with parathyroidectomy. Clinical and biochemical evaluation is performed at the inclusion, and 6, 12, 36 and 60 months. A biocollection is collected. The main hypotheses are that parathyroidectomy could improve cardiovascular, renal, bone, and cardiovascular outcomes along with quality of life.

DETAILED DESCRIPTION:
Primaty hyperparathyroidism is the third most frequent endocrine disorder, which only curative treatment is the parathyroidectomy (approximately 8000/year). However, evidences suggest that the mildest forms of PHPT could be safely monitored with simple surveillance. However, to define surgical indications is challenging because data regarding the impach of surgery on several outcomes (namely cardiovascular, bone, renal or quality of life) are controversial.

CoHPT is a prospective, monocentric, observational cohort including all consecutive patients diagnosed with sporadic primary hyperparathyroidism in Nantes University Hospital aiming to study the outcomes associated with parathyroidectomy. Patients are followed even if surgery is not performed.

A systematic clinical and biochemical evaluation is performed at the inclusion, and 6, 12, 36 and 60 months. These informations include demographic and general medical data, pre-operative imaging exams, post-operative outcomes, histopathological analysis, evaluation of the impact of primary hyperparathyroidism and its surgery on target organs (bone, kidney, cardiovascular) and quality of life. Fasting blood samples are also collected to constitute a biocollection, in order to measure biomarkers related to the bone remodeling and the cardiovascular risk.

The objectives are:

* To know the long-term consequences of the primary hyperparathyroidism treatment or observation.
* To better define the surgical indications
* To better understand the mechanisms of the cardiovascular impairment by using the biocollection
* To study the medico-economics consequences of the surgical management versus simple surveillance

ELIGIBILITY:
Inclusion Criteria:

• Age > 18

Exclusion Criteria:

* Age < 18
* Pregnancy / lactation
* Adults underguardianship
* Secondary/tertiary hyperparathyroidism
* Multiple endocrine neoplasia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients consulting for sporadic primary hyperparathyroidism in Nantes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 403 (Estimated)
Dates: Start 2016-03-31 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2027-02-24 (Estimated)

PRIMARY OUTCOMES:
Occurrence of cardiovascular events, after parathyroidectomy for primary hyperparathyroidism | Between inclusion and 12 months after surgery
  Cardiovascular events include myocardial infarction, cerebrovascular and peripheral arterial events
Change in LDL-cholesterol concentration after surgery | Between inclusion and 12 months after surgery
  Plasma LDL-cholesterol (mg/dL) will be directly measured using enzymatic method
Change in HDL-cholesterol concentration after surgery | Between inclusion and 12 months after surgery
  Plasma HDL-cholesterol (mg/dL) will be measured using enzymatic method
Change in plasma triglycerides concentration after surgery | Between inclusion and 12 months after surgery
  Plasma triglycerides (mg/dL) will be measured using enzymatic method
Change in homeostasis model assessment HOMA-IR index after surgery | Between inclusion and 12 months after surgery
  HOMA-IR is calculated using fasting plasma glucose and insulin level, with the following formula: (fasting plasma insulin (mIU/L) × fasting plasma glucose (mmol/L))/22.5
Change in homeostasis model assessment HOMA-B index after surgery | Between inclusion and 12 months after surgery
  HOMA-B is calculated using fasting plasma glucose and insulin level, with the following formula: 20 × fasting plasma insulin (mIU/L)/[fasting plasma glucose (mmol/L) - 3.5]
Change in arterial stiffness after surgery | Between inclusion and 12 months after surgery
  Arterial stiffness is reflected by the measurement of the pulse wave velocity using the PoPmeter® instrument

SECONDARY OUTCOMES:
Occurrence of cardiovascular events, after parathyroidectomy for primary hyperparathyroidism | Between inclusion and 60 months after surgery
  Cardiovascular events include myocardial infarction, cerebrovascular and peripheral arterial events
Change in LDL-cholesterol concentration after surgery | Between inclusion and 60 months after surgery
  Plasma LDL-cholesterol (mg/dL) will be directly measured using enzymatic method
Change in HDL-cholesterol concentration after surgery | Between inclusion and 60 months after surgery
  Plasma HDL-cholesterol (mg/dL) will be measured using enzymatic method
Change in plasma triglycerides concentration after surgery | Between inclusion and 60 months after surgery
  Plasma triglycerides (mg/dL) will be measured using enzymatic method
Change in homeostasis model assessment HOMA-IR index after surgery | Between inclusion and 60 months after surgery
  HOMA-IR is calculated using fasting plasma glucose and insulin level, with the following formula: (fasting plasma insulin (mIU/L) × fasting plasma glucose (mmol/L))/22.5
Change in homeostasis model assessment HOMA-B index after surgery | Between inclusion and 60 months after surgery
  HOMA-B is calculated using fasting plasma glucose and insulin level, with the following formula: 20 × fasting plasma insulin (mIU/L)/[fasting plasma glucose (mmol/L) - 3.5]
Change in arterial stiffness after surgery | Between inclusion and 60 months after surgery
  Arterial stiffness is reflected by the measurement of the pulse wave velocity using the PoPmeter® instrument
Change in bone mineral density after parathyroidectomy | Between inclusion and 12 months after surgery
  Bone mineral density is measured using Dual X-ray absorptiometry on lumbar spine, left hip, left femoral neck and left distal radius
Change in bone-specific alkaline phosphatases | Between inclusion and 12 months after surgery
  Alkaline phosphatases (IU/L) are measured using ELISA enzymatic method
Change in P1NP | Between inclusion and 12 months after surgery
  P1NP (µg/L) are measured using ELISA enzymatic method
Change in plasma CTX | Between inclusion and 12 months after surgery
  CTX (µg/L) are measured using ELISA enzymatic method
Change in bone mineral density after parathyroidectomy | Between inclusion and 60 months after surgery
  Bone mineral density is measured using Dual X-ray absorptiometry on lumbar spine, left hip, left femoral neck and left distal radius
Change in bone-specific alkaline phosphatases | Between inclusion and 60 months after surgery
  Alkaline phosphatases (IU/L) are measured using ELISA enzymatic method
Change in P1NP | Between inclusion and 60 months after surgery
  P1NP (µg/L) are measured using ELISA enzymatic method
Change in plasma CTX | Between inclusion and 60 months after surgery
  CTX (µg/L) are measured using ELISA enzymatic method
Change in the physical component score of the SF-36 questionnaire after surgery | Between inclusion and 36 months after surgery
  The physical component score is calculated from 4 items of the SF-36 questionnaire related to physical health. Results are expressed as a ratio between the included patients with values expected in an age- and sex-matched French reference population (available in Perneger T, Leplège A, Ecosse E. Le questionnaire MOS SF-36: manuel de l'utilisateur et guide d'interprétation des scores; Paris: Editions Estem. 2001:1-156.)
Change in the mental component score of the SF-36 questionnaire after surgery | Between inclusion and 36 months after surgery
  The mental component score is calculated from 4 items of the SF-36 questionnaire related to mental health. Results are expressed as a ratio between the included patients with values expected in an age- and sex-matched French reference population.
Change in the physical component score of the SF-36 questionnaire after surgery | Between inclusion and 60 months after surgery
  The physical component score is calculated from 4 items of the SF-36 questionnaire related to physical health. Results are expressed as a ratio between the included patients with values expected in an age- and sex-matched French reference population (available in Perneger T, Leplège A, Ecosse E. Le questionnaire MOS SF-36: manuel de l'utilisateur et guide d'interprétation des scores; Paris: Editions Estem. 2001:1-156.)
Change in the mental component score of the SF-36 questionnaire after surgery | Between inclusion and 60 months after surgery
  The mental component score is calculated from 4 items of the SF-36 questionnaire related to mental health. Results are expressed as a ratio between the included patients with values expected in an age- and sex-matched French reference population.
Change in renal outcomes (estimated glomerular filtration rate) after parathyroidectomy | Between inclusion and 60 months after surgery
  Estimated glomerular filtration rate will be calculated using the CKD-EPI equation from the measured serum creatinine
Medico-economic impact of parathyroidectomy for primary hyperparathyroidism in comparison with simple surveillance | 60 months after surgery
  Takes into account the incidence of the worsening of cardiac and bone comorbidities and surgical complications. Data will be cross-referenced by probabilistic matching with the data of the Système National d'Information Interrégimes d'Assurance Maladie (SNIIR-AM)

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loison M, Wargny M, Caillard C, Guillot P, Le Bras M, Cariou B, Blanchard C, Mirallie E, Frey S. Radius Bone Mineral Density Measurement Is Essential During Initial PHPT Workup: Results of a Retrospective Study on 400 Patients. World J Surg. 2026 Jan 4. doi: 10.1002/wjs.70223. Online ahead of print. PMID 41486083
- [Derived] Frey S, Perrot B, Caillard C, Le Bras M, Gerard M, Blanchard C, Cariou B, Wargny M, Mirallie E. Parathyroidectomy for primary hyperparathyroidism: effect on quality of life after 3 years - a prospective cohort study. Int J Surg. 2023 Mar 1;109(3):364-373. doi: 10.1097/JS9.0000000000000282. PMID 36917123